CLINICAL TRIAL: NCT06870110
Title: Brain Training for Substance Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurotype Inc. (Industry)
Collaborators: University of Minnesota (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071720; R43DA057773-01A1 (NIH); R44DA059517-01 (NIH)
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
Keywords: biofeedback; neurofeedback; electroencephalogram; addiction; substance use disorder; opioid use disorder; attention; emotion regulation; event-related potential
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Substance-Related Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Biofeedback (Experimental)
  Interventions: Device: Bias Modification Biofeedback

INTERVENTIONS:
Device: Bias Modification Biofeedback — The device uses EEG-based bias modification biofeedback intended to reduce attention to drug-related cues and increase attention to non-drug pleasant scenes. Specifically, the device measures perceptual biases from Event-Related Potential biomarkers related to Substance Use Disorders.
  Other Names: Modit™; Modit-O™; Modit-AB™

SUMMARY:
Participants play games designed to train visual attention towards natural, non-drug-related scenarios. A biofeedback loop between gameplay and an electroencephalogram (EEG) system monitors game performance and guides game difficulty.

DETAILED DESCRIPTION:
The main purpose of this project is to gather pilot data on neurofeedback games that use electroencephalogram (EEG)-based Attention Bias Modification (ABM) to reduce cue-induced drug craving processes in individuals with Opioid Use Disorder (OUD). The project will involve the use of three empirically-supported and potentially therapeutic games that include drug- (such as pill bottle and syringe) and non-drug-related stimuli (such as food and smiling faces). An EEG system will be used to monitor brain activity during gameplay.

The neurofeedback loop for attention training will be synchronized to cue presentations using EEGs which monitor visual Event-Related Potentials (ERP) signatures of attention. The degree of difficulty (i.e., cue content) on subsequent trials of the game will be determined based on the level of attention measured in the neurofeedback loop.

ELIGIBILITY:
Inclusion Criteria:

OUD patient participants:

* Admitted into chemical treatment with opioid use being a reason for treatment;
* DSM-IV-TR diagnosis of OUD;
* Ability to provide informed consent;
* A minimum of a 6th grade reading level; and
* Able and willing to provide own contact information for follow-up visit(s).

Control participants:

* Age- and gender-matched to an OUD patient participant in the study;
* Ability to provide informed consent;
* A minimum of a 6th grade reading level;
* Able and willing to provide own contact information for follow-up visit(s).

Exclusion Criteria:

OUD patient participants:

* Refusal or inability to consent;
* Pregnant;
* History of serious neurological illness (e.g., Chronic seizure disorder, Wernicke-Korsakoff Syndrome, Epilepsy, Any history of seizures not caused by withdrawal from substances, Other [please specify]);
* Inability to see text and photos clearly on the computer display; and
* Unwillingness to change hairstyle (e.g., braids, pony tails, dreadlocks) or remove wig to accommodate application of the EEG headset, if necessary.

Control participants:

* Refusal or inability to consent;
* Pregnant;
* History of serious neurological illness (e.g., Chronic seizure disorder, Wernicke-Korsakoff Syndrome, Epilepsy, Any history of seizures, Other [please specify]);
* Inability to see text and photos clearly on the computer display;
* Current or previous problems using opioids, other prescription (prescribed or not prescribed) or illicit drugs;
* Regular nicotine user (e.g., cigarette smoker, e-cig user) within the past 12 months; and
* Unwillingness to change hairstyle (e.g., braids, pony tails, dreadlocks) or remove wig to accommodate application of the EEG headset, if necessary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in ERP-Based Classification of Opioid-Related Attention Bias (Probability Score) | Pre- to post-biofeedback session (same day, approximately 30 minutes)
  The primary outcome will be the change in ERP-based classification scores (probability values) reflecting opioid-related attention bias. ERP voltages from all electrodes will be classified with coefficients reflecting increased amplitude in Early Posterior Negativity (150 to 300 ms), P300 complex (250 to 450 ms), and Late Positive Potential (400 to 900 ms) windows. Change in classification score from the last minus first block will be evaluated.
Change in Visual Probe Task Reaction Time (milliseconds) to Drug-Related Stimuli | Pre- to post-biofeedback session (same day, approximately 30 minutes)
  The primary outcome will be the change in reaction time (milliseconds) on the Visual Probe Task, measuring attention bias toward drug-related versus neutral stimuli. Participants will complete the task before and after the biofeedback session. Attention bias is indicated by differences in reaction time when responding to probes replacing drug-related versus neutral stimuli. Improvement is reflected by reduced bias scores, calculated as the difference between reaction times to drug-related versus neutral probes. Change scores from pre- to post-session will be analyzed.

SECONDARY OUTCOMES:
Change in Rating of Cue Reactivity (1-5 Likert Scale) | Pre- to post-biofeedback for a given scene (same day, approximately 30 seconds)
  The outcome will be the change in self-reported cue reactivity, measured with a Likert scale ranging from 1 (not at all) to 5 (extremely). Participants rate their cue reactivity before and after each series of images being presented for a given scene. The average change in cue reactivity across all scenes during the 30-minute biofeedback protocol will be quantified for each session.
Change in Visual Analog Scale (VAS) Rating of Instantaneous Opioid Craving (1-100) | Pre- to post-biofeedback session (same day, approximately 30 minutes)
  The outcome will be the change in self-reported instantaneous ("right now") opioid craving, measured with a Visual Analog Scale (VAS) ranging from 1 ("No Drug Craving") to 100 ("Extreme Drug Craving"). Participants will rate their current craving before and after the biofeedback session. Change scores from pre- to post-session will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Anker, PhD, Principal Investigator — University of Minnesota; Scott Burwell, PhD, Study Director — Neurotype Inc.
Locations (1):
- University of Minnesota - Department of Psychiatry & Behavioral Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared upon request based on decision of study leadership.